CLINICAL TRIAL: NCT04065893
Title: Impact of Catheter Ablation of Ventricular Arrhythmias on Suboptimal Biventricular Pacing in Cardiac Resynchronization Therapy
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Other Study IDs: CRT-Bivent.
Record Dates: First submitted 2019-08-16; First posted 2019-08-22 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Systolic Heart Failure; Ventricular Premature Complexes; Ventricular Tachycardia; Cardiac Resynchronization Therapy; Reduced Biventricular Pacing
MeSH Terms: conditions — Heart Failure, Systolic; Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Catheter ablation group: Patients with reduced biventricular pacing due to PVC or VT receiving catheter ablation of PVC/VT according to guidelines and clinical practices
  Interventions: Procedure: Catheter ablation of ventricular arrhythmia
- Medical treatment group: Patients with reduced biventricular pacing due to PVC or VT receiving intensified medical therapy (antiarrhythmics/betablocker) according to guidelines and clinical practices
  Interventions: Drug: Intensified medical therapy

INTERVENTIONS:
Procedure: Catheter ablation of ventricular arrhythmia — PVC or VT ablation
  Groups: Catheter ablation group
Drug: Intensified medical therapy — Dosage increase / new onset of Betablocker / medical antiarrhythmic medication according to guideline and clinical practice
  Groups: Medical treatment group

SUMMARY:
Cardiac resynchronization therapy reduces mortality in patients with systolic heart failure and left bundle branch block. Reduced biventricular pacing can lead to therapy failure. Most effective mortality reduction was seen with a BiV pacing above 98%.

Reduced BiV pacing is a common phenomenon with potential impact on CRT-response and pts' prognosis. Frequent ventricular ectopy may be associated with attenuated benefit from CRT. The investigators sought to systematically assess the effect of ventricular arrhythmia treatment on BiV pacing.

ELIGIBILITY:
Inclusion Criteria:

* reduced biventricular pacing <98% due to ventricular arrhythmia

Exclusion Criteria:

* reduced biventricular pacing <98% due to other cause
* age <18
* pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pts. with systolic heart failure, wide QRS complex and CRT with reduced biventricular pacing due to ventricular arrhythmia (PVC/VT)
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Biventricular pacing | 3 month after intervention biventricular pacing (%) is routinely monitored
  Influence of intervention (Ablation/medical treatment) on previously reduced biventricular pacing percentage (<98%). Biventricular pacing is measured in percentage of stimulation and is monitored at routine device interrogation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Bruck JH, Middeldorp M, Sultan A, Scheurlen C, Seuthe K, Wormann J, Filipovic K, Kadhim K, Sanders P, Steven D, Luker J. Impact of ventricular arrhythmia management on suboptimal biventricular pacing in cardiac resynchronization therapy. J Interv Card Electrophysiol. 2023 Mar;66(2):353-361. doi: 10.1007/s10840-022-01259-0. Epub 2022 Jun 14. PMID 35697890